CLINICAL TRIAL: NCT06235073
Title: Robotic and Manual Cochlear Implantation: An Intra-individual Study of Speech Recognition and Electrode Holder Position
Brief Title: Robotic and Manual Cochlear Implantation: An Intra-individual Study of Speech Recognition and Electrode Holder Position (ICRobMan)
Acronym: ICRobMan
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0107 - ICRobMan
Record Dates: First submitted 2023-10-19; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-10

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Manual implantation
- Robot assisted implantation

SUMMARY:
Cochlear implantation (CI) allows rehabilitation for patients with severe to profound hearing impairment. Although the use of a robotic assistant provides technical assistance to the surgeon, the assessment of the impact of its use on auditory outcomes remains uncertain, due to inter-individual variability of preoperative audiometric thresholds and the various possible intrascalar positions of the electrode array. WThe investigators aim to compare the hearing results of patients who underwent bilateral cochlear implantation, one side was performed with manual insertion and the other side with robot-assisted insertion. The electrode array intrascalar positioning and the surgery duration were also studied.

This retrospective intra-individual study involved 10 patients who underwent bilateral cochlear implantation. The unique composition of this cohort enabled the investigators to utilize each patient as their own control.

DETAILED DESCRIPTION:
Cochlear implantation (CI) allows rehabilitation for patients with severe to profound hearing impairment. Although the use of a robotic assistant provides technical assistance to the surgeon, the assessment of the impact of its use on auditory outcomes remains uncertain, due to inter-individual variability of preoperative audiometric thresholds and the various possible intrascalar positions of the electrode array. The investigators aim to compare the hearing results of patients who underwent bilateral cochlear implantation, one side was performed with manual insertion and the other side with robot-assisted insertion. The electrode array intrascalar positioning and the surgery duration were also studied.

This retrospective intra-individual study involved 10 patients who underwent bilateral cochlear implantation. The unique composition of this cohort enabled the investigators to utilize each patient as their own control.

ELIGIBILITY:
Inclusion Criteria:

* bilateral cochlear implantation at a tertiary referral center
* one side manual
* one side robot-assisted

Exclusion Criteria:

* opposition
* under curatorship

Ages: 44 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective intra-individual study involved 10 patients who underwent bilateral cochlear implantation at a tertiary referral center. Manual cochlear implantations were performed between January 2006 and June 2020, while robot-assisted implantations took place between September 2020 and May 2022. Sequential implantation was applied to 9 of the patients, while 1 patient underwent both manual and robot-assisted cochlear implantations in a single procedure.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Speech disyllabic recognition | at 1 year

SECONDARY OUTCOMES:
Pure tone average | At 1 year
Intrascalar positionning | Postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Chru de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement